CLINICAL TRIAL: NCT01834365
Title: Effect of Structured Education to Decrease Blood Pressure for Hypertension in Elderly : a Randomized Controlled Trial
Brief Title: Effect of Structured Education to Decrease Blood Pressure for Hypertension in Elderly
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Ayatullah Khomaini, MD, Effect of Structured Education to Decrease Blood Pressure for Hypertension in Elderly : a randomized controlled trial, Indonesia University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: AKhomaini
Record Dates: First submitted 2013-04-10; First posted 2013-04-17 (Estimated); Last update posted 2013-04-17 (Estimated); Status verified 2013-04

CONDITIONS: Hypertension
Keywords: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Checklist

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Structured education & checklist (Experimental): Formatted education and checklist every month for 3 months
  Interventions: Other: Structured education; Other: Checklist
- Structured education (Active Comparator): Formatted education every month for 3 months
  Interventions: Other: Structured education
- Without Structured Education with checklist (Active Comparator): No structured education with checklist
  Interventions: Other: Without structure education with checklist

INTERVENTIONS:
Other: Structured education — Formatted education about hypertension
  Arms: Structured education; Structured education & checklist
Other: Checklist
  Arms: Structured education & checklist
Other: Without structure education with checklist
  Arms: Without Structured Education with checklist

SUMMARY:
There is a structured educational effect on blood pressure reduction in elderly hypertensive patients.

DETAILED DESCRIPTION:
Eligibility criteria are men and women over 60 years old and available to participate in the study for 3 months with blood pressure higher than 140/90.

Exclusion criteria are severe dementia, malignant hypertension, depression

Outcome measures are systolic and diastolic blood pressure after 3 months administration of structured education once a month.

ELIGIBILITY:
Inclusion Criteria:

* Subject with age more than 60 years
* Blood pressure higher than 140/90

Exclusion Criteria:

* Severe Dementia
* Depression
* Malignant Hypertension

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-10; Primary Completion 2013-02 (Actual); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure | 3 Months
  We aim to measure the difference in systolic blood pressure after 3 months administration structured education in elderly with hypertension

SECONDARY OUTCOMES:
Diastolic blood pressure | 3 Months
  We measure the difference of diastolic blood pressure after 3 Months administration of structured education in elderly with hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Ayatullah Khomaini, MD, Principal Investigator — Faculty of Medicine University of Indonesia
Locations (1):
- Cipto Mangunkusumo National Hospital Recruiting, Jakarta, Indonesia